CLINICAL TRIAL: NCT00295243
Title: A Phase I Trial of the Dual Kinase Inhibitor GW572016 in Combination With Topotecan in Patients With Advanced Solid Malignancies
Brief Title: Phase I Study of GW572016 With Topotecan to Treat Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Julian R. Molina, M.D., Ph.D., Mayo Clinic Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1073-04; MC0315 (Other: Mayo Clinic Cancer Center); 1073-04 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Advanced Solid Malignancies
MeSH Terms: interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan

SUMMARY:
Participants will take GW572016 by mouth daily each cycle (cycles 28 days in length) and will be given Topotecan intravenously on Days 1, 8 and 15.

DETAILED DESCRIPTION:
Participants will take GW572016 by mouth daily each cycle (cycles 28 days in length) and will be given Topotecan intravenously on Days 1, 8 and 15. During Cycle 1 participants will be required to spend the evening before Day 1 in the General Clinical Research Center and frequent blood samples will be drawn on Day 1; this schedule will be repeated the evening of Day 6 with the blood samples drawn on Day 7. Participants will have weekly CBCs.

ELIGIBILITY:
Age 18 and older Histologic proof of cancer that is unresectable ANC greater than 1500 u/L PLC greater than 100,000 u/L Total bilirubin less then or equal to ULN AST less than 3 x ULN or AST less than 5 x ULN if liver involvement Creatinine less than 1.5 x ULN Hemoglobin greater than 9 g/dL Echocardiogram with ejection fraction great than 40% Life expectancy of more than 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
find the highest dose of GW572016 and Topotecan that can be safely given together
Learn the side effects of GW572016 and Topotecan when given together
Learn whether GW572016 changes how the body handles or processesTopotecan
Learn whether Topotecan changes how the body handles or processes GW572016

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States